CLINICAL TRIAL: NCT02772172
Title: Accuracy of Dental Implant Placement Using Two Different CBCT-derived Templates: a Randomized Controlled Clinical Trial
Brief Title: Accuracy of Dental Implant Placement Using Two Different CBCT-derived Templates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhuofan Chen, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZhuofanChen
Record Dates: First submitted 2016-05-04; First posted 2016-05-13 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-05

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GuideMia surgical template (Active Comparator): A radiographic guide is prepared before CT/CBCT scan. The CT/CBCT scan DICOM ﬁles are loaded in GuideMia program and converted into 3D computer images. A surgical template is fabricated through this virtual planning.
  Interventions: Device: Surgical Template
- Control surgical template (Active Comparator): A radiographic guide is prepared before CT/CBCT scan. The CT/CBCT scan DICOM ﬁles are loaded in control program and converted into 3D computer images. A surgical template is fabricated through this virtual planning.
  Interventions: Device: Surgical Template

INTERVENTIONS:
Device: Surgical Template
  Other Names: GuideMia; control

SUMMARY:
The main purpose of the present study is to evaluate the dental implant placement using two different CBCT-derived templates and to study the related factors that affect accuracy so as to support the further clinical application of the technique. Thirty patients with partial edentulous denture are recruited. They are randomized to two groups. A radiographic guide is prepared before CT/CBCT scan. The CT/CBCT scan DICOM ﬁles are loaded in a planning program and converted into 3D computer images. A surgical template is fabricated through this virtual planning. After 6 weeks, if the implants are judged stable, the patient has the option of replacing the ﬁxed prosthesis. Patients are recalled for oral hygiene maintenance and prosthetic controls every 6 months for the entire duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Partial edentulism
* Missing more than three teeth in succession
* Presence of adjacent teeth
* Systemically healthy
* Good maxillomandibular relation
* Maximal mouth opening>5 mm

Exclusion Criteria:

* Poor oral hygiene
* Severe parafunctional habits, for example, bruxing and clenching
* Presence of clinically active periodontal disease as expressed by probing pocket depths≥4 mm in combination with bleeding on probing
* Maxillary sinus involvement
* Conditions that might lead to a possibly lowered regenerative capacity of the bone, for example, osteoporosis and Paget's disease
* Pregnant or expecting to be pregnant
* History of drug and alcohol abuse
* History of systemic diseases that would contraindicate oral surgical treatment, for example, uncontrolled diabetes (defined as HBA1c level >7%)
* Radiotherapy in the head and neck area
* On certain medications like bisphosphonates or steroids currently or within the past three months
* Unwillingness to return for the follow-up examination
* Smokers (more than20 cigarettes per day). Subjects smoking <20 cigarettes per day were requested to stop smoking before and after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-11 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Position changes between the planned and achieved implant position | Change from preoperative to postoperative within 1 week
  Accuracy analysis. The linear and angular deviations between the planned and achieved implant position are analyzed.

SECONDARY OUTCOMES:
Implant and prosthesis survival | Up to 18 months after baseline
  Implant and prosthesis survival will be determined at 6 months，12months and 18 months
Radiographic bone level | Up to 18 months after baseline
  Radiographic bone level will be recorded at 6 months，12months and 18 months
The incidence of biological and mechanical complications | Up to 18 months after baseline
  The incidence of biological and mechanical complications will be recorded at baseline, 6 months，12months and 18 months
Probing depth | Up to 18 months after baseline
  Probing depth will be recorded at 6 months，12months and 18 months
Modified plaque index | Up to 18 months after baseline
  Modified plaque index will be recorded at 6 months，12months and 18 months
Modified bleeding index | Up to 18 months after baseline
  Modified bleeding index will be recorded at 6 months，12months and 18 months
Gingival index | Up to 18 months after baseline
  Gingival index will be recorded at 6 months，12months and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhuofan Chen, professor, Principal Investigator — School of Stomatology, Hospital of Stomatology, Sun Yat-Sen University
Locations (1):
- Guanghua school of stomatology, hospital of stomtology, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lopes A, Malo P, de Araujo Nobre M, Sanchez-Fernandez E. The NobelGuide(R) All-on-4(R) Treatment Concept for Rehabilitation of Edentulous Jaws: A Prospective Report on Medium- and Long-Term Outcomes. Clin Implant Dent Relat Res. 2015 Oct;17 Suppl 2:e406-16. doi: 10.1111/cid.12260. Epub 2014 Sep 5. PMID 25195544
- [Result] Sun Y, Luebbers HT, Agbaje JO, Schepers S, Politis C, Van Slycke S, Vrielinck L. Accuracy of Dental Implant Placement Using CBCT-Derived Mucosa-Supported Stereolithographic Template. Clin Implant Dent Relat Res. 2015 Oct;17(5):862-70. doi: 10.1111/cid.12189. Epub 2013 Dec 16. PMID 24341829
- [Result] Polizzi G, Cantoni T. Five-year follow-up of immediate fixed restorations of maxillary implants inserted in both fresh extraction and healed sites using the NobelGuide system. Clin Implant Dent Relat Res. 2015 Apr;17(2):221-33. doi: 10.1111/cid.12102. Epub 2013 Jun 23. PMID 23789721